CLINICAL TRIAL: NCT06736665
Title: Comparative Efficacy of Orbital Atherectomy and Intravascular Lithotripsy in the Treatment of Calcified Coronary Nodules. The ORBIT-SHOCK Pilot Study.
Brief Title: Orbital Atherectomy vs Intravascular Lithotripsy for the Treatment of Calcified Coronary Nodules (ORBIT-SHOCK).
Acronym: ORBIT-SHOCK
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Luis Manuel Domínguez Rodríguez, Interventional Cardiologist and Clinical Researcher, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORBIT-SHOCK
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Coronary Arterial Disease (CAD); Coronary Calcification; Coronary Calcified Nodules; Orbital Atherectomy; Intravascular Lithotripsy; Optical Coherence Tomography (OCT); Percutaneous Coronary Intervention (PCI); Chronic Coronary Syndrome; Acute Coronary Syndrome (ACS)
Keywords: Coronary arterial disease; Coronary calcification; Coronary calcified nodules; Orbital atherectomy; Intravascular lithotripsy; Optical Coherence Tomography (OCT); Percutaneous Coronary Intervention (PCI); Chronic Coronary Syndrome; Acute Coronary Syndrome (ACS); ORBIT-SHOCK; ORBIT SHOCK
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Tomography, Optical Coherence; Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Once the presence of a calcified nodular lesion is confirmed and the patient meets the inclusion criteria without any exclusion criteria, the patient will be randomized to one of the two treatment techniques being evaluated in the study (OA vs. IVL) in a 1:1 ratio. A stratified randomization will be implemented based on the type of calcified nodule (eruptive or non-eruptive) to ensure equal proportions of each type between the two treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Orbital atherectomy (Active Comparator): The Diamondback-360 (OAS) (Abbott) device is used to perform this technique, consisting of a bidirectional, diamond-coated orbital crown that utilizes a combination of centrifugal force (creating elliptical orbits) and surface abrasion to modify the calcified plaque and increase distensibility. Additionally, the pulsatile impact of the crown at high speed can create microfractures in deep calcium. As a result, a single 1.25 mm crown can treat vessels ranging from 2.5 to 4 mm in diameter.
  Interventions: Device: Orbital atherectomy; Device: Optical Coherence Tomography (OCT); Device: Percutaneous coronary intervention with stent implantation
- Intravascular lithotripsy (Active Comparator): The Shockwave Medical Intravascular Lithotripsy System (Shockwave Medical) is a balloon that emits pulsatile sonic waves capable of fracturing intracoronary calcium. This therapy is administered by advancing a catheter and inflating the balloon at low pressure to deliver sonic pulses.
  Interventions: Device: Intravascular lithotripsy; Device: Optical Coherence Tomography (OCT); Device: Percutaneous coronary intervention with stent implantation

INTERVENTIONS:
Device: Orbital atherectomy — The Diamondback-360 (OAS) (Abbott) device is used to perform this technique, consisting of a bidirectional, diamond-coated orbital crown that utilizes a combination of centrifugal force (creating elliptical orbits) and surface abrasion to modify the calcified plaque and increase distensibility. Additionally, the pulsatile impact of the crown at high speed can create microfractures in deep calcium. As a result, a single 1.25 mm crown can treat vessels ranging from 2.5 to 4 mm in diameter.
  Arms: Orbital atherectomy
Device: Intravascular lithotripsy — The Shockwave Medical Intravascular Lithotripsy System (Shockwave Medical) is a balloon that emits pulsatile sonic waves capable of fracturing intracoronary calcium. This therapy is administered by advancing a catheter and inflating the balloon at low pressure to deliver sonic pulses.
  Other Names: Shockwave
  Arms: Intravascular lithotripsy
Device: Optical Coherence Tomography (OCT) — Optical Coherence Tomography (OCT) is an intravascular imaging modality that uses near-infrared light to provide high-definition, cross-sectional and three-dimensional images of the vessel microstructure.
  These images provide additional information on the degree and characteristics of coronary artery disease compared to angiography which doesn't delineate the composition of the coronary artery. With automated, highly accurate measurements, OCT can guide stent selection, placement, and deployment.
Device: Percutaneous coronary intervention with stent implantation — All patients will undergo percutaneous coronary intervention with drug-eluting stent implantation after plaque modification using the technique assigned by randomization.

SUMMARY:
The ORBIT-SHOCK pilot study is a multicenter, prospective, randomized clinical trial initiated by investigators. It will include patients diagnosed with atherosclerotic coronary artery disease presenting calcified nodules (CN), identified by optical coherence tomography (OCT), causing significant angiographic stenosis and eligible for revascularization through percutaneous coronary intervention (PCI).

Patients will be randomized in a 1:1 ratio to undergo lesion preparation with either orbital atherectomy (OA) or intravascular lithotripsy (IVL).

The ORBIT-SHOCK pilot study is a multicenter, prospective, randomized clinical trial initiated by investigators. It will include patients diagnosed with atherosclerotic coronary artery disease presenting calcified nodules (CN), identified by optical coherence tomography (OCT), causing significant angiographic stenosis and eligible for revascularization through percutaneous coronary intervention (PCI). Patients will be randomized in a 1:1 ratio to undergo lesion preparation with either orbital atherectomy (OA) or intravascular lithotripsy (IVL).

The aim of this pilot trial is to compare PCI outcomes and the incidence of adverse events between both techniques.

DETAILED DESCRIPTION:
Coronary calcification in the form of calcified nodules (CN) is systematically associated with worse outcomes due to the difficulty in adequately dilation of the lesion and the inability to properly fracture the calcium nodule before stent implantation.

The ORBIT-SHOCK pilot study is a multicenter, prospective, randomized clinical trial initiated by investigators. It will include patients diagnosed with atherosclerotic coronary artery disease presenting CNs, identified by optical coherence tomography (OCT), causing significant angiographic stenosis and eligible for revascularization through percutaneous coronary intervention (PCI).

Patients will be randomized in a 1:1 ratio to undergo lesion preparation with either orbital atherectomy (OA) or intravascular lithotripsy (IVL).

Primary endpoint: Compare both techniques in terms of achieving adequate stent expansion, measured by OCT.

Secondary endpoints: Evaluate procedural and strategy success rates, assess their impact on calcium nodule modification, and monitor the incidence of adverse clinical events at 12 months.

Patients will be monitored for 12 months after the procedure to assess the incidence of adverse events during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years.
2. Atherosclerotic coronary artery disease with calcified nodules identified by OCT in a native vessel, eligible for percutaneous coronary revascularization.
3. Clinical presentation of chronic coronary syndrome or acute coronary syndrome without ST elevation*.
4. Distal vessel reference diameters ≥ 2.5 mm and ≤ 4.0 mm. * Non-culprit lesions eligible for revascularization in a staged procedure following a ST-elevation myocardial infarction (STEMI) are considered for inclusion.

Exclusion Criteria:

1. Culprit lesions in acute coronary syndrome with ST elevation.
2. Left main disease.
3. In-stent restenosis lesions.
4. Critical stenoses where it is not possible to advance the OCT catheter across the lesion after predilation with a balloon of up to 2 mm in diameter.
5. Lesion involving a bifurcation with a secondary branch diameter ≥2 mm.
6. Cardiogenic shock.
7. Patients requiring cardiac surgery or percutaneous valve intervention within three months before or after angioplasty.
8. Pregnancy.
9. Life expectancy of less than one year.
10. Contraindication for the use of appropriate antiplatelet therapy post-revascularization.
11. Coronary artery disease with an indication for surgical revascularization.
12. Advanced chronic kidney disease or anatomical characteristics that contraindicate the use of optical coherence tomography.
13. Inability to obtain informed consent.
14. Allergy to eggs or soy, contraindicating the use of OA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stent expansion | At the end of percutaneous coronary intervention
  Percentage of stent expansion at the CN site: measured with OCT, defined as the ratio between the minimum stent area at the CN site and the average of the distal and proximal reference areas.

SECONDARY OUTCOMES:
Procedural success | At the end of percutaneous coronary intervention
  Achieving a stent expansion of ≥ 80% with TIMI III flow, in the absence of stent loss, coronary perforation, or intraprocedural death.
Strategy success | At the end of percutaneous coronary intervention
  Defined as procedural success without the need for crossover to an alternative treatment.
Minimum stent area | At the end of percutaneous coronary intervention
  Minimum stent area (MSA)
Minimum stent area at the CN site. | At the end of percutaneous coronary intervention
  Minimum stent area at the CN site.
Significant stent malapposition at the CN site | At the end of percutaneous coronary intervention
  Measured using OCT, defined as a stent strut detachment ≥ 0.4 mm from the underlying vessel wall, with a longitudinal extension ≥ 1 mm.
Degree of calcium nodule debulking | At the end of percutaneous coronary intervention
  Reduction in calcium nodule size (mm²), measured after plaque modification and prior to stent implantation.
Evidence of fracture at the CN site | At the end of percutaneous coronary intervention
  Evidence of new disruption or discontinuity observed on OCT after plaque modification and prior to stent implantation.
Degree of stent ellipticity at the CN site | At the end of percutaneous coronary intervention
  Measured using OCT at the end of the procedure, calculated as the ratio of the maximum luminal diameter to the minimum luminal diameter of the stent at the CN site.
Residual luminal protrusion of the calcium nodule following stent implantation | At the end of percutaneous coronary intervention
  Residual luminal protrusion of the calcium nodule following stent implantation, measured by OCT in mm2.
Target lesion failure (TLF) at 12 months | At 12 months
  Composite of clinically driven target lesion revascularization, myocardial infarction or cardiac death related to the target lesion.
Target lesion revascularization (TLR) at 12 months | At 12 months
  Repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Major Adverse Cardiovascular Events (MACE) at 12 months | At 12 months
  Defined as a composite of cardiovascular death, non-fatal target lesion myocardial infarction, unplanned target lesion revascularization or stent thrombosis.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario General de Alicante, Alicante
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Result] Lansky AJ, Messe SR, Brickman AM, Dwyer M, van der Worp HB, Lazar RM, Pietras CG, Abrams KJ, McFadden E, Petersen NH, Browndyke J, Prendergast B, Ng VG, Cutlip DE, Kapadia S, Krucoff MW, Linke A, Moy CS, Schofer J, van Es GA, Virmani R, Popma J, Parides MK, Kodali S, Bilello M, Zivadinov R, Akar J, Furie KL, Gress D, Voros S, Moses J, Greer D, Forrest JK, Holmes D, Kappetein AP, Mack M, Baumbach A. Proposed Standardized Neurological Endpoints for Cardiovascular Clinical Trials: An Academic Research Consortium Initiative. J Am Coll Cardiol. 2017 Feb 14;69(6):679-691. doi: 10.1016/j.jacc.2016.11.045. PMID 28183511
- [Result] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; ESC Scientific Document Group. Fourth universal definition of myocardial infarction (2018). Eur Heart J. 2019 Jan 14;40(3):237-269. doi: 10.1093/eurheartj/ehy462. No abstract available. PMID 30165617
- [Result] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Eur Heart J. 2018 Jun 14;39(23):2192-2207. doi: 10.1093/eurheartj/ehy223. PMID 29897428
- [Result] Maehara A, Ben-Yehuda O, Ali Z, Wijns W, Bezerra HG, Shite J, Genereux P, Nichols M, Jenkins P, Witzenbichler B, Mintz GS, Stone GW. Comparison of Stent Expansion Guided by Optical Coherence Tomography Versus Intravascular Ultrasound: The ILUMIEN II Study (Observational Study of Optical Coherence Tomography [OCT] in Patients Undergoing Fractional Flow Reserve [FFR] and Percutaneous Coronary Intervention). JACC Cardiovasc Interv. 2015 Nov;8(13):1704-14. doi: 10.1016/j.jcin.2015.07.024. PMID 26585621
- [Result] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Result] Holm NR, Andreasen LD, Neghabat O, Laanmets P, Kumsars I, Bennett J, Olsen NT, Odenstedt J, Hoffmann P, Dens J, Chowdhary S, O'Kane P, Bulow Rasmussen SH, Heigert M, Havndrup O, Van Kuijk JP, Biscaglia S, Mogensen LJH, Henareh L, Burzotta F, H Eek C, Mylotte D, Llinas MS, Koltowski L, Knaapen P, Calic S, Witt N, Santos-Pardo I, Watkins S, Lonborg J, Kristensen AT, Jensen LO, Calais F, Cockburn J, McNeice A, Kajander OA, Heestermans T, Kische S, Eftekhari A, Spratt JC, Christiansen EH; OCTOBER Trial Group. OCT or Angiography Guidance for PCI in Complex Bifurcation Lesions. N Engl J Med. 2023 Oct 19;389(16):1477-1487. doi: 10.1056/NEJMoa2307770. Epub 2023 Aug 27. PMID 37634149
- [Result] Ali ZA, Landmesser U, Maehara A, Matsumura M, Shlofmitz RA, Guagliumi G, Price MJ, Hill JM, Akasaka T, Prati F, Bezerra HG, Wijns W, Leistner D, Canova P, Alfonso F, Fabbiocchi F, Dogan O, McGreevy RJ, McNutt RW, Nie H, Buccola J, West NEJ, Stone GW; ILUMIEN IV Investigators. Optical Coherence Tomography-Guided versus Angiography-Guided PCI. N Engl J Med. 2023 Oct 19;389(16):1466-1476. doi: 10.1056/NEJMoa2305861. Epub 2023 Aug 27. PMID 37634188
- [Result] Lee JM, Choi KH, Song YB, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Jeong JO, Song PS, Doh JH, Jo SH, Yoon CH, Kang MG, Koh JS, Lee KY, Lim YH, Cho YH, Cho JM, Jang WJ, Chun KJ, Hong D, Park TK, Yang JH, Choi SH, Gwon HC, Hahn JY; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging-Guided or Angiography-Guided Complex PCI. N Engl J Med. 2023 May 4;388(18):1668-1679. doi: 10.1056/NEJMoa2216607. Epub 2023 Mar 5. PMID 36876735
- [Result] Shin D, Dakroub A, Singh M, Malik S, Sakai K, Maehara A, Shlofmitz E, Jeremias A, Shlofmitz RA, Ali ZA. Debulking Effect of Orbital Atherectomy for Calcified Nodule Assessed by Optical Coherence Tomography. Circ Cardiovasc Interv. 2024 Aug;17(8):e014145. doi: 10.1161/CIRCINTERVENTIONS.124.014145. Epub 2024 Jul 1. No abstract available. PMID 38946577
- [Result] Chiang CSM, Alan Chan KC, Lee M, Chan KT. Orbital-Tripsy: Novel Combination of Orbital-Atherectomy and Intravascular-Lithotripsy, in Calcified Coronaries After Failed Intravascular-Lithotripsy. JACC Case Rep. 2020 Dec 16;2(15):2437-2444. doi: 10.1016/j.jaccas.2020.10.027. eCollection 2020 Dec. PMID 34317190
- [Result] Rola P, Wlodarczak S, Barycki M, Furtan L, Jastrzebski A, Kedzierska M, Doroszko A, Lesiak M, Wlodarczak A. Safety and Efficacy of Orbital Atherectomy in the All-Comer Population: Mid-Term Results of the Lower Silesian Orbital Atherectomy Registry (LOAR). J Clin Med. 2023 Sep 8;12(18):5842. doi: 10.3390/jcm12185842. PMID 37762782
- [Result] Okamoto N, Ueda H, Bhatheja S, Vengrenyuk Y, Aquino M, Rabiei S, Barman N, Kapur V, Hasan C, Mehran R, Baber U, Kini AS, Sharma SK. Procedural and one-year outcomes of patients treated with orbital and rotational atherectomy with mechanistic insights from optical coherence tomography. EuroIntervention. 2019 Apr 20;14(17):1760-1767. doi: 10.4244/EIJ-D-17-01060. PMID 29957595
- [Result] Yamamoto MH, Maehara A, Karimi Galougahi K, Mintz GS, Parviz Y, Kim SS, Koyama K, Amemiya K, Kim SY, Ishida M, Losquadro M, Kirtane AJ, Haag E, Sosa FA, Stone GW, Moses JW, Ochiai M, Shlofmitz RA, Ali ZA. Mechanisms of Orbital Versus Rotational Atherectomy Plaque Modification in Severely Calcified Lesions Assessed by Optical Coherence Tomography. JACC Cardiovasc Interv. 2017 Dec 26;10(24):2584-2586. doi: 10.1016/j.jcin.2017.09.031. No abstract available. PMID 29268891
- [Result] Yamamoto MH, Maehara A, Kim SS, Koyama K, Kim SY, Ishida M, Fujino A, Haag ES, Alexandru D, Jeremias A, Sosa FA, Karimi Galougahi K, Kirtane AJ, Moses JW, Ali ZA, Mintz GS, Shlofmitz RA. Effect of orbital atherectomy in calcified coronary artery lesions as assessed by optical coherence tomography. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):1211-1218. doi: 10.1002/ccd.27902. Epub 2018 Oct 17. PMID 30328257
- [Result] Okamoto N, Egami Y, Nohara H, Kawanami S, Sugae H, Kawamura A, Ukita K, Matsuhiro Y, Nakamura H, Yasumoto K, Tsuda M, Matsunaga-Lee Y, Yano M, Nishino M, Tanouchi J. Direct Comparison of Rotational vs Orbital Atherectomy for Calcified Lesions Guided by Optical Coherence Tomography. JACC Cardiovasc Interv. 2023 Sep 11;16(17):2125-2136. doi: 10.1016/j.jcin.2023.06.016. PMID 37704299
- [Result] Faria D, Vinhas H, Bispo J, Guedes J, Marto S, Palmeiro H, Franco P, Mimoso J. Initial experience with orbital atherectomy in a non-surgical center in Portugal. Rev Port Cardiol. 2024 Dec;43(12):659-665. doi: 10.1016/j.repc.2024.03.005. Epub 2024 Jul 8. English, Portuguese. PMID 38986811
- [Result] Florek K, Bartoszewska E, Biegala S, Klimek O, Malcharczyk B, Kubler P. Rotational Atherectomy, Orbital Atherectomy, and Intravascular Lithotripsy Comparison for Calcified Coronary Lesions. J Clin Med. 2023 Nov 23;12(23):7246. doi: 10.3390/jcm12237246. PMID 38068298
- [Result] Chambers JW, Feldman RL, Himmelstein SI, Bhatheja R, Villa AE, Strickman NE, Shlofmitz RA, Dulas DD, Arab D, Khanna PK, Lee AC, Ghali MG, Shah RR, Davis TP, Kim CY, Tai Z, Patel KC, Puma JA, Makam P, Bertolet BD, Nseir GY. Pivotal trial to evaluate the safety and efficacy of the orbital atherectomy system in treating de novo, severely calcified coronary lesions (ORBIT II). JACC Cardiovasc Interv. 2014 May;7(5):510-8. doi: 10.1016/j.jcin.2014.01.158. PMID 24852804
- [Result] Parikh K, Chandra P, Choksi N, Khanna P, Chambers J. Safety and feasibility of orbital atherectomy for the treatment of calcified coronary lesions: the ORBIT I trial. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1134-9. doi: 10.1002/ccd.24700. Epub 2013 Mar 5. PMID 23460596
- [Result] Ali ZA, Kereiakes D, Hill J, Saito S, Di Mario C, Honton B, Gonzalo N, Riley R, Maehara A, Matsumura M, Stone GW, Shlofmitz R. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Calcified Nodules. JACC Cardiovasc Interv. 2023 May 8;16(9):1122-1124. doi: 10.1016/j.jcin.2023.02.015. Epub 2023 Apr 5. No abstract available. PMID 37029020
- [Result] Akasaka T, Kubo T. OCT-derived coronary calcified nodules as a predictor of high-risk patients. EuroIntervention. 2020 Aug 28;16(5):361-363. doi: 10.4244/EIJV16I5A65. No abstract available. PMID 32855116
- [Result] Prati F, Gatto L, Fabbiocchi F, Vergallo R, Paoletti G, Ruscica G, Marco V, Romagnoli E, Boi A, Fineschi M, Calligaris G, Tamburino C, Crea F, Ozaki Y, Alfonso F, Arbustini E. Clinical outcomes of calcified nodules detected by optical coherence tomography: a sub-analysis of the CLIMA study. EuroIntervention. 2020 Aug 28;16(5):380-386. doi: 10.4244/EIJ-D-19-01120. PMID 32310133
- [Result] Ali ZA, Kereiakes DJ, Hill JM, Saito S, Di Mario C, Honton B, Gonzalo N, Riley RF, Maehara A, Matsumura M, Shin D, Stone GW, Shlofmitz RA. Impact of Calcium Eccentricity on the Safety and Effectiveness of Coronary Intravascular Lithotripsy: Pooled Analysis From the Disrupt CAD Studies. Circ Cardiovasc Interv. 2023 Oct;16(10):e012898. doi: 10.1161/CIRCINTERVENTIONS.123.012898. Epub 2023 Oct 17. PMID 37847770
- [Result] McInerney A, Travieso A, Jeronimo Baza A, Alfonso F, Del Val D, Cerrato E, Garcia de Lara J, Pinar E, Perez de Prado A, Jimenez Quevedo P, Tirado-Conte G, Nombela-Franco L, Brugaletta S, Cepas-Guillen P, Sabate M, Cubero Gallego H, Vaquerizo B, Jurado A, Varbella F, Jimenez M, Garcia Escobar A, de la Torre JM, Amat Santos I, Jimenez Diaz VA, Escaned J, Gonzalo N. Impact of coronary calcium morphology on intravascular lithotripsy. EuroIntervention. 2024 May 20;20(10):e656-e668. doi: 10.4244/EIJ-D-23-00605. PMID 38776142
- [Result] Brott BC. The Calcified Nodule Paradox. JACC Cardiovasc Interv. 2023 May 8;16(9):1036-1038. doi: 10.1016/j.jcin.2023.04.001. No abstract available. PMID 37164600
- [Result] Sato T, Matsumura M, Yamamoto K, Shlofmitz E, Moses JW, Khalique OK, Thomas SV, Tsoulios A, Cohen DJ, Mintz GS, Shlofmitz RA, Jeremias A, Ali ZA, Maehara A. Impact of Eruptive vs Noneruptive Calcified Nodule Morphology on Acute and Long-Term Outcomes After Stenting. JACC Cardiovasc Interv. 2023 May 8;16(9):1024-1035. doi: 10.1016/j.jcin.2023.03.009. PMID 37164599